CLINICAL TRIAL: NCT01904682
Title: A Single-arm Study to Assess the Efficacy and Safety of Oral Rigosertib in Transfusion-dependent, Low or Intermediate-1, Myelodysplastic Syndrome Patients Based on the International Prognostic Scoring System
Brief Title: Oral Rigosertib in Low Risk MDS Patients Refractory to ESAs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 09-07; 2013-000672-15 (EudraCT Number)
Record Dates: First submitted 2013-07-14; First posted 2013-07-22 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: Erythrocyte transfusion; Erythropoiesis-stimulating agent; International Prognostic Scoring System
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral rigosertib (Experimental): Patients will take 560 mg oral rigosertib (two 280 mg capsules) in the morning and 280 mg (one 280 mg capsule) in the afternoon, in fasting conditions, for 21 consecutive days of 21-day cycle (continuous regimen).
  Interventions: Drug: Oral rigosertib

INTERVENTIONS:
Drug: Oral rigosertib — Dose of 560 mg consists of two (2) 280 mg soft gel capsules of rigosertib.
  Other Names: ON 01910.Na; rigosertib sodium

SUMMARY:
The study will enroll low risk MDS patients who need red blood cell transfusions and who are refractory to or are not using erythropoiesis-stimulating agents. The purpose of the study is to determine whether oral rigosertib treatment results in hematological improvements according to the 2006 International Working Group criteria in these patients. The study will also record any side effects that may occur during the study.

DETAILED DESCRIPTION:
This will be a Phase II, single-arm, multicenter study (approximately 15 centers). Approximately 40 transfusion-dependent patients with Low- or Int-1 risk Myelodysplastic Syndrome (MDS) by International Prognostic Scoring System (IPSS) will be enrolled and treated with oral rigosertib administered twice daily for 21 consecutive days of a 21-day cycle (continuous regimen) in order to obtain at least 35 evaluable patients treated for at least 8 weeks. Patients will take 560 mg rigosertib (two 280 mg capsules) in the morning and 280 mg (one 280 mg capsule) in the afternoon, in fasting conditions. All patients on intermittent regimen at the time of Amendment 2 of the Protocol will be switched to the continuous regimen, including patients on reduced doses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS according to World Health Organization (WHO) criteria (Appendix 2) or French-American-British (FAB) classification that must be confirmed by bone marrow (BM) aspirate and/or biopsy within 6 weeks prior to Screening.
* Myelodysplastic syndrome (MDS) classified as Low risk or Int-1 risk, according to International Prognostic Scoring System (IPSS) classification; in addition, patients should never have been classified as Int-2 or High-risk since their MDS was diagnosed;
* Transfusion dependency defined by transfusion of at least 4 units of Red blood cells (RBC) within 56 days before Screening (pre-transfusion Hgb values values must be ≤ 9 g/dL to be taken into account).
* Refractory to 8- to 12-week course of Erythropoiesis-stimulating agent (ESA) administered within the past 2 years before enrollment, or erythropoietin (EPO) level ˃ 500 mU/mL and off ESA for at least 8 weeks before Screening.
* Off all other treatments for MDS (azacitidine, decitabine, lenalidomide, chemotherapy, immunotherapy) for at least 2 weeks prior to Screening.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0, 1 or 2.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* The patient must signed an informed consent form (ICF) indicating that s/he understands the purpose of, and procedures required for, the study and is willing to participate.

Exclusion Criteria:

* Ongoing clinically significant anemia due to factors such as iron, vitamin B12, or folate deficiencies, auto-immune or hereditary hemolysis, or gastrointestinal (GI) bleeding.
* Serum ferritin < 50 ng/mL.
* Hypoplastic MDS (cellularity <10%)
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin ≥ 2.0 mg/dL not related to hemolysis or Gilbert's disease.
* Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 2.5 x the upper limit of normal (ULN).
* Serum creatinine ≥ 2.0 mg/dL.
* Ascites requiring active medical management including paracentesis.
* Hyponatremia (defined as serum sodium value of < 130 mEq/L).
* Female patients who are pregnant or lactating.
* Patients of childbearing potential who are unwilling to follow strict contraception requirements.
* Female patients with reproductive potential who do not have a negative blood or urine pregnancy test at Screening.
* Major surgery without full recovery or major surgery within 3 weeks of Screening.
* Uncontrolled hypertension (defined as a systolic pressure ≥ 160 mmHg and/or a diastolic pressure ≥ 110 mmHg).
* New onset seizures (within 3 months prior to the first dose of rigosertib) or poorly controlled seizures.
* Any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy.
* Chronic use (˃ 2 weeks) of corticosteroids (˃ 10 mg/24 hr equivalent prednisone) within 4 weeks of Screening.
* Investigational therapy within 4 weeks of Screening.
* Allergy to a local anaesthetic.
* Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07; Primary Completion 2020-12 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Hematologic Improvement | 24 Weeks
  The number of patients who achieve hematologic improvement will be documented. Hematologic improvement is defined by the 2006 International Working Group (IWG) response criteria for the erythroid, platelet and neutrophil lineages.

SECONDARY OUTCOMES:
Overall Response | Up to 2 years
  The number of patients with a complete remission or a partial remission will be documented. Complete remission and partial remission are defined according to 2006 IWG response criteria for MDS. Overall response = complete remission + partial remission.
Duration of Response | Up to 2 years
  The number of weeks a complete remission or a partial remission is observed in a patient will be documented.
Number of Adverse Events | Up to 2 years
  Specific safety parameters and procedures will include recording of medical history, medication history, physical examination, measurement of vital signs (blood pressure, temperature, respiration rate, and pulse), weight, laboratory evaluations, and toxicity and AE assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Fruchtman, MD, Study Chair — Traws Pharma, Inc.
Locations (14):
- United States (10):
  - Stanford University School of Medicine, Stanford, California
  - Anschutz Cancer Pavilion University of Colorado, Aurora, Colorado
  - Washington Cancer Institute at Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - The University of Chicago, Chicago, Illinois
  - Greenbaum Cancer Center University of Maryland, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Hôpital Saint-Louis, Service d'Hématologie, Paris, IDF, France
- Germany (3):
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Heinrich Heine Universität, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony

REFERENCES:
- [Background] Seetharam M, Fan AC, Tran M, Xu L, Renschler JP, Felsher DW, Sridhar K, Wilhelm F, Greenberg PL. Treatment of higher risk myelodysplastic syndrome patients unresponsive to hypomethylating agents with ON 01910.Na. Leuk Res. 2012 Jan;36(1):98-103. doi: 10.1016/j.leukres.2011.08.022. Epub 2011 Sep 14. PMID 21924492
- [Background] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.